CLINICAL TRIAL: NCT00695955
Title: A One-Year Phase 3, Open-Label Study to Evaluate the Safety and Tolerability of TAK-491 in Subjects With Essential Hypertension
Brief Title: One-Year Safety and Tolerability Study of Azilsartan Medoxomil in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 01-05-TL-491-006; U1111-1113-8874 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Essential Hypertension; Cardiovascular Disease; High Blood Pressure; Drug Therapy
MeSH Terms: conditions — Hypertension; Essential Hypertension; Cardiovascular Diseases | interventions — azilsartan medoxomil; azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azilsartan Medoxomil (Experimental)
  Interventions: Drug: Azilsartan medoxomil with or without add-on chlorthalidone; Drug: Azilsartan medoxomil with or without add-on hydrochlorothiazide

INTERVENTIONS:
Drug: Azilsartan medoxomil with or without add-on chlorthalidone — Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks; increased to azilsartan medoxomil 80 mg, tablets, orally, once daily for remainder of 56-week treatment period, if tolerated. Additional antihypertensive medications added, beginning with chlorthalidone 25 mg, once-daily, if target blood pressure not achieved.
  Other Names: TAK-491; Edarbi
Drug: Azilsartan medoxomil with or without add-on hydrochlorothiazide — Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks; increased to azilsartan medoxomil 80 mg, tablets, orally, once daily for remainder of 56-week treatment period, if tolerated. Additional antihypertensive medications added, beginning with hydrochlorothiazide 12.5 to 25 mg, once-daily, if target blood pressure not achieved.
  Other Names: TAK-491; Edarbi

SUMMARY:
This purpose of this study is to evaluate the long-term safety and tolerability of azilsartan medoxomil in individuals with essential hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive treatments, hypertension remains inadequately controlled; only about one-third of patients continue to maintain control successfully.

Takeda Global Research and Development is developing TAK-491 (azilsartan medoxomil) for the treatment of essential hypertension. This study is being conducted to demonstrate the long-term safety and tolerability of azilsartan medoxomil in individuals with essential hypertension.

Study participation is anticipated to be approximately 1 year and 1.5 months, and participants will be required to return to the clinic for 10 study visits.

ELIGIBILITY:
Inclusion Criteria

1. Diastolic blood pressure greater than or equal to 95 mm Hg and less than or equal to 119 mm Hg. For diabetic subjects and subjects with chronic kidney disease, diastolic blood pressure must be greater than or equal to 85 mm Hg and less than or equal to109 mm Hg).
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating.
3. Clinical laboratory evaluations within the reference range for or deemed not clinically significant by the investigator.

Exclusion Criteria

1. Systolic blood pressure greater than 185 mm Hg.
2. Expected to take angiotensin II receptor blockers other than the study drug.
3. Taking more than 2 antihypertensive agents.
4. Hypersensitive to angiotensin II receptor blockers, thiazide-type diuretics or sulfonamide-derived compounds.
5. Recent history of major cardiovascular event.
6. History of moderate to severe heart failure or hypertensive encephalopathy.
7. Clinically significant cardiac conduction defects.
8. Secondary hypertension of any etiology.
9. Known or suspected unilateral or bilateral renal artery stenosis.
10. Severe renal dysfunction or disease.
11. History of drug abuse or a history of alcohol abuse within the past 2 years.
12. Previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug..
13. Uncontrolled diabetes mellitus.
14. Alanine aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
15. Serum potassium level of greater than the upper limit of normal.
16. Currently is participating in another investigational study or has participated in an investigational study within 30 days prior to enrollment.
17. Any other serious disease or condition.
18. Randomized in a previous azilsartan medoxomil study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (41):
- United States (39):
  - Ozark, Alabama
  - Tallassee, Alabama
  - Long Beach, California
  - Santa Rosa, California
  - Spring Valley, California
  - Colorado Springs, Colorado
  - Trumbull, Connecticut
  - Waterbury, Connecticut
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Brooklyn Center, Minnesota
  - Olive Branch, Mississippi
  - Rochester, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Mogadore, Ohio
  - Springdale, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Anderson, South Carolina
  - Mt. Pleasant, South Carolina
  - Simpsonville, South Carolina
  - Bristol, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - North Richland Hills, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
- San Bernardo, Santiago Metropolitan, Chile
- Tijuana, Estado de Baja California, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 39 investigative sites in Chile, Mexico and the United States from 22 June 2007 to 30 April 2010.
Pre-assignment Details: Participants with essential hypertension were enrolled in a once-daily (QD) treatment group.
Groups:
- Azilsartan Medoxomil: Cohort 1: Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks; increased to azilsartan medoxomil 80 mg, tablets, orally, once daily for remainder of 56-week treatment period, if tolerated. Additional antihypertensive medications added, beginning with chlorthalidone 25 mg, once-daily, if target blood pressure not achieved.
  Cohort 2: Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks; increased to azilsartan medoxomil 80 mg, tablets, orally, once daily for remainder of 56-week treatment period, if tolerated. Additional antihypertensive medications added, beginning with hydrochlorothiazide 12.5 to 25 mg, once-daily, if target blood pressure not achieved.
Period: Cohort 1
Arm/Group | Azilsartan Medoxomil
Started | 362
Completed | 260
Not Completed | 102
Not completed — Adverse Event | 26
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 30
Not completed — Withdrawal by Subject | 25
Not completed — Lack of Efficacy | 3
Not completed — Other | 16
Period: Cohort 2
Arm/Group | Azilsartan Medoxomil
Started | 307
Completed | 203
Not Completed | 104
Not completed — Adverse Event | 24
Not completed — Protocol Violation | 5
Not completed — Lost to Follow-up | 38
Not completed — Withdrawal by Subject | 28
Not completed — Lack of Efficacy | 4
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Azilsartan Medoxomil
Number analyzed (Participants) | 669
Age, Customized [Number; unit: participants]
  <45 years (Cohort 1) | 81
  Between 45 and 64 years (Cohort 1) | 233
  ≥65 years (Cohort 1) | 48
  <45 years (Cohort 2) | 90
  Between 45 and 64 years (Cohort 2) | 193
  ≥65 years (Cohort 2) | 24
Sex/Gender, Customized [Number; unit: participants]
  Female (Cohort 1) | 173
  Male (Cohort 1) | 189
  Female (Cohort 2) | 144
  Male (Cohort 2) | 163

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events From Day 1 Through End of the Study - Cohort 1.
Description: Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after the last dose of study drug, or if a serious adverse event, within 30 days after the last dose of study drug.
Time Frame: 56 weeks.
Population: Full Analysis Set.
Measure: Number; unit: participants
Groups:
- Cohort 1: Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks; increased to azilsartan medoxomil 80 mg, tablets, orally, once daily for remainder of 56-week treatment period, if tolerated. Additional antihypertensive medications added, beginning with chlorthalidone 25 mg, once-daily, if target blood pressure not achieved.
Arm/Group | Cohort 1
Number analyzed (Participants) | 362
participants
  Number of Participants | 267
  Percentage of Participants | 73.8

2. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events From Day 1 Through End of the Study - Cohort 2.
Description: as for outcome 1
Time Frame: 56 weeks.
Population: Full Analysis Set.
Measure: Number; unit: participants
Groups:
- Cohort 2: Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks; increased to azilsartan medoxomil 80 mg, tablets, orally, once daily for remainder of 56-week treatment period, if tolerated. Additional antihypertensive medications added, beginning with hydrochlorothiazide 12.5 to 25 mg, once-daily, if target blood pressure not achieved.
Arm/Group | Cohort 2
Number analyzed (Participants) | 307
participants
  Number of Participants | 241
  Percentage of Participants | 78.5

3. Secondary Outcome: Change From Baseline in Sitting Clinic Systolic Blood Pressure - Cohort 1.
Description: The change between sitting clinic systolic blood pressure measured at each week assessed relative to the baseline measurement. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Time Frame: 52 weeks
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1
Number analyzed (Participants) | 362
mmHg
  Week 4 | -10.1 (15.21)
  Week 8 | -13.1 (16.72)
  Week 12 | -21.5 (15.80)
  Week 16 | -25.4 (15.09)
  Week 26 | -26.3 (15.97)
  Week 36 | -27.3 (16.63)
  Week 46 | -28.1 (17.21)
  Week 56 | -25.2 (18.05)
  Final Visit | -22.1 (18.64)

4. Secondary Outcome: Change From Baseline in Sitting Clinic Systolic Blood Pressure - Cohort 2
Description: as for outcome 3
Time Frame: 52 weeks
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 2
Number analyzed (Participants) | 307
mmHg
  Week 4 | -14.4 (13.57)
  Week 8 | -17.5 (15.07)
  Week 12 | -23.8 (15.97)
  Week 16 | -26.2 (15.65)
  Week 26 | -24.8 (15.25)
  Week 36 | -22.5 (14.89)
  Week 46 | -23.8 (15.35)
  Week 56 | -24.2 (15.96)
  Final Visit | -22.7 (17.14)

5. Secondary Outcome: Change From Baseline in Sitting Clinic Diastolic Blood Pressure - Cohort 1.
Description: The change between sitting clinic diastolic blood pressure measured at each week assessed relative to the baseline measurement. Mean calculated by using the average (arithmetic mean) of 3 measurements performed at each visit.
Time Frame: 52 weeks.
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 1
Number analyzed (Participants) | 362
mmHg
  Week 4 | -8.9 (8.73)
  Week 8 | -11.0 (9.97)
  Week 12 | -15.9 (9.12)
  Week 16 | -18.7 (9.06)
  Week 26 | -18.6 (9.15)
  Week 36 | -19.9 (9.13)
  Week 46 | -19.8 (9.67)
  Week 56 | -18.4 (9.52)
  Final Visit | -16.5 (10.23)

6. Secondary Outcome: Change From Baseline in Sitting Clinic Diastolic Blood Pressure - Cohort 2.
Description: as for outcome 5
Time Frame: 52 weeks.
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cohort 2
Number analyzed (Participants) | 307
mmHg
  Week 4 | -10.6 (9.23)
  Week 8 | -12.3 (9.05)
  Week 12 | -16.8 (9.48)
  Week 16 | -18.2 (10.28)
  Week 26 | -17.7 (10.95)
  Week 36 | -16.2 (9.08)
  Week 46 | -17.2 (9.57)
  Week 56 | -17.9 (10.85)
  Final Visit | -16.2 (11.05)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) defined as any AEs, regardless of relationship to study drug, that occur after the first dose of study drug and within 14 days after last dose, or if an SAE, within 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 30/362 | 22/307
Other Adverse Events (participants affected / at risk) | 134/362 | 106/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=362) | Cohort 2 (N=307)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Maculopathy (Eye disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Splenic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope vasovagal (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=362) | Cohort 2 (N=307)
Dizziness (Nervous system disorders) | 52 | 44
Headache (Nervous system disorders) | 38 | 28
Fatigue (General disorders) | 32 | 16
Upper respiratory tract infection (Infections and infestations) | 25 | 20
Urinary tract infection (Infections and infestations) | 26 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.